CLINICAL TRIAL: NCT02493283
Title: Pharmacokinetics and Distribution of Dapsone (DDS) in Leucocytes After Single-dose and Multiple-dose Administration in Healthy Subjects Genotyped for CYP2C9 and NAT2 and in Patients With Autoimmune Bullous Dermatoses
Brief Title: Pharmacokinetics and Distribution of Dapsone in Leucocytes After Single-dose and Multiple-dose Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Dapson - 2010
Record Dates: First submitted 2015-06-30; First posted 2015-07-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Methemoglobinemia; Linear IgA Bullous Dermatosis
Keywords: dapsone; blood leucocytes; pharmacokinetics; metabolism
MeSH Terms: conditions — Methemoglobinemia; Linear IgA Bullous Dermatosis | interventions — Dapsone; Leukocyte Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment A (Active Comparator): single-dose administration of 100 mg dapsone; sampling of blood, urine and feces; sampling for leucocytes collection and sampling for additional safety analyses (Met-Hb)
  Interventions: Drug: Dapsone single dose; Biological: leucocytes; Biological: Met-Hb
- Treatment B (Active Comparator): multiple-dose administration of 100 mg dapsone s.i.d. for 7 days; sampling of blood, urine and feces; sampling for leucocytes collection and sampling for additional safety analyses (Met-Hb)
  Interventions: Drug: Dapsone multiple dose; Biological: leucocytes; Biological: Met-Hb

INTERVENTIONS:
Drug: Dapsone single dose — Administration of two tablets Dapson-Fatol 50 mg Tabletten (= 100 mg dapsone) and sampling of blood (before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 h after single-dose administration), urine (0-24 h, 24-48 h, 48-72 h, 72-96 h, 96 -120 h) and feces (on treatment days 1-5)
  Arms: Treatment A
Drug: Dapsone multiple dose — Administration of two tablets Dapson-Fatol 50 mg Tabletten (= 100 mg dapsone) s.i.d. for 7 days and sampling of blood (before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 h after last repeated-dose administration), urine (last treatment day 0-24 h) and feces (on treatment days 12-15)
  Arms: Treatment B
Biological: leucocytes — sampling for leucocytes collection: study days -1, 1, 14 and 15
Biological: Met-Hb — sampling before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 h after single-dose administration, before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 h after last repeated-dose administration and sampling for additional safety analyses (Met-Hb): study days 10, 12, 14 and hematology on study day 12

SUMMARY:
The objectives of the study are

* to evaluate pharmacokinetics, distribution in blood leucocytes, metabolism and methemoglobinemia after single-dose and repeated-dose administration of 100 mg of dapsone in healthy subjects genotyped for CYP2C9 and NAT2
* to evaluate serum through levels, distribution in blood leucocytes and methemoglobinemia after repeated-dose treatment with dapsone in patients with autoimmune bullous dermatoses before and after concomitant treatment with glucocorticoids

DETAILED DESCRIPTION:
Dapsone (diamino diphenyl sulphone, DDS) was synthesized by Emil Fromm and Jakob Wittmann in Freiburg (Germany) in 1908. In 1937, the anti-inflammatory potency of dapsone was discovered in experimentally-induced infections in mice. Since 1941, dapsone (as Promin®) is used with great success in the therapy of leprosy. Dapsone is a mainstay in the treatment of leprosy, being one of the components of the multidrug regimen advised by the World Health Organization (WHO).

In 1950, Esteves and Brandão confirmed the efficacy of the drug in patients with dermatitis herpetiformis Duhring. Sneddon and Wilkinson in England reported a remission as caused by dapsone in a patient with subcorneal pustulosis. The efficacy of dapsone in treatment of pemphigus vulgaris was initially reported by Winkelmann and Roth in 1960.

After oral administration, dapsone is almost completely absorbed from the gastrointestinal tract with bioavailability of more than 86 %. Maximum serum concentrations between 0,63 and 4,82 mg/l are attained within 2-8 hours after single doses between 50 mg and 300 mg. At steady-state, the serum concentration fluctuate between 3,26 mg/l and 1,95 mg/l chronic treatment with 100 mg dapsone once daily (s.i.d.).

Dapsone is distributed to all organs, it crosses the blood-brain barrier and placenta and is detected in breast milk.

About 20% of dapsone is excreted unchanged into the urine, 70-85% as water-soluble metabolites additionally to a small amount in feces.

Dapsone is nearly completely metabolized in the liver and in activated polymorphic neutrophils (PMN) and/or mononuclear cells. The major metabolic pathway in the liver is N-acetylation by the polymorphic N-acetyltransferase 2 (NAT2) and N-oxidation by cytochrome P-450 (CYP) enzymes. Major metabolites are monoacetyl-dapsone (MADDS) and dapsone hydroxylamine (DDS-NOH). Dapsone undergoes enterohepatic circulation.

MADDS is subjected also to significant deacetylation. A constant equilibrium between acetylation and deacetylation is reached within a few hours after the oral administration of either dapsone or MADDS. The acetylation ratio shows a large interindividual variation, ranging from 0.1 to 2.0. These ratios show a bimodal distribution pattern.

Acetylation is not the rate-determining step in overall elimination of dapsone. The amount of MADDS excreted in urine is very low because it is largely deacetylated to dapsone before excretion into the urine. Between slow acetylators (SA) and rapid acetylators (RA), there are no differences neither in dapsone serum concentrations nor any pharmacokinetic parameters of dapsone. Also, the therapeutic response is the same in both acetylator phenotypes.

However, excretion of both MADDS and its conjugated derivatives is higher in RA. Therefore, dapsone may be used for determination of the NAT2 phenotype even though these metabolites represent only a very small fraction of the dose.

MADDS is highly bound to plasma proteins (> 98%), about 20-25 times more tightly than dapsone. Presumably, the small fraction of unbound MADDS and its strong binding to plasma proteins are reasons for its low availability in erythrocytes (erythrocyte/plasma ratio = 0.33). Tight protein binding is also the reason behind low glomerular filtration rate of the metabolite; therefore the half-life for MADDS is approximately 20-25 hours, similar like for dapsone.

Microsomal N-hydoxylation is the second major metabolic route of dapsone which seems to be associated with hematological side effects of the drug. However, the data on excretion of free and conjugated DDS-NOH vary widely in the literature. No reliable information is available on excretion of hydroxylated MADDS compounds.

In terms of efficacy and safety of dapsone, most important is the generation of DDS-NOH, that also occurs in inflamed lesions of the skin as mediated by activated PMN. Thus, over the years, dapsone became a first-line drug in the treatment of dermatitis herpetiformis Duhring, Sneddon-Wilkinson-Syndrome and further bullous autoimmune dermatoses. Most recently was found, that formation of DDS-NOH is mainly under control of CYP2C9 in-vitro.(Lit.) Because of the known CYP2C9 gene polymorphisms (about 4-6 % are poor metabolizers, PM), efficacy of the drug in bullous autoimmune dermatoses may be dependent on the metabolizer status of the patients.

The investigators hypothesize, that subjects which are slow acetylators of NAT2 (SA) but extensive metabolizers of CYP2C9 (EM) may form significantly higher levels of the active metabolite DDS-NOH than rapid acetylators of NAT2 (RA) being PM of CYP2C9 (PM).

ELIGIBILITY:
Inclusion Criteria:

* 18 - 45 years
* preferably males (females will be included if there are not enough males which fulfill the inclusion criteria)
* Caucasian
* body weight: > 19 kg/m² and < 27 kg/m²
* good health as evidenced by the results of the clinical examination, ECG, and the laboratory check-up, which are judged by the clinical investigator not to differ in a clinical relevant way from the normal state
* written informed consent given by volunteer after being provided with detailed information about the nature, risks, and scope of the clinical trial as well as the expected desirable and adverse effects of the drug

Exclusion Criteria:

* results of the medical examination or laboratory screening which are judged by the clinical investigator to differ in a clinically relevant way from the normal state
* female subjects not willing to apply a highly effective method of birth control, which means contraceptive methods with a low failure rate of less than 1% per year during the entire study as stated in the Note for Guidance on Non-Clinical Safety Studies for the Conduct of Human Clinical Trials for Pharmaceuticals (CPMP/ICH/286/95, modifications). These methods include implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner.
* subjects with existing cardiac or hematological diseases and/ or pathological findings which might interfere with safety, pharmacodynamic effect and/ or pharmacokinetics of dapsone
* subjects with existing gastrointestinal diseases and/ or pathological findings which might interfere with safety, pharmacodynamic effect and/ or pharmacokinetics of dapsone
* subjects with acute or chronic organ diseases which could affect drug absorption, metabolism or excretion of dapsone and its metabolites
* subjects liable to orthostatic dysregulation, fainting, or blackout
* subjects with known allergic reactions to the investigational product and its adjuvants
* deficiency of glucose-6-phosphate dehydrogenase (G6PD)
* subjects positive of HBsAG, HIV and /or drugs
* subjects with history of psychiatric disorders (depressions, other psychotic disorders)
* subjects with history of epilepsy
* gravidity
* breast feeding mothers, lactation
* alcohol consumption more than 20 g/day
* special or uniform nutritional habits, e.g. vegetarians or undercaloric diet
* intake of grapefruit containing food or beverages and poppy seeds containing products (will not be allowed) 14 days prior to the first drug administration (and) until the last blood sampling of the study
* subjects with uncommon physical exercise (competitive athletes), excessive physical activity one week before the trial
* excessive smoking (more than 10 cigarettes or equivalents per day)
* less than 14 days after last acute disease
* less than 14 days after last systemic or local drug administration or less than 10 half-lives of the respective drugs
* blood donation within the last 3 months
* blocking time due to another clinical trial with investigational products
* subjects suspected or known not to follow instructions
* subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to as a result of their participation in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) for dapsone (DDS) and MA-DDS | before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours after single-dose administration and before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours after last repeated-dose administration
  AUC0-∞ for single dose administration and AUC0-24h for multiple dose

SECONDARY OUTCOMES:
maximal serum concentration (Cmax) for dapsone (DDS) and MA-DDS | before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours after single-dose administration and before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours after last repeated-dose administration
minimal serum concentration (Cmin) for dapsone (DDS) and MA-DDS | before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours after last repeated-dose administration on study-day 15
peak trough fluctuation (PTF) for dapsone (DDS) and MA-DDS | before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours after last repeated-dose administration on study-day 15
timepoint of maximal serum concentration (Tmax) for dapsone (DDS) and MA-DDS | before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours after single -dose administration and before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours after last repeated-dose administration
terminal half live (T1/2) for dapsone (DDS) and MA-DDS | before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours after single-dose administration and before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours after last repeated-dose administration
renal clearance (CLR) for dapsone (DDS) and MA-DDS | before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96 and 120 hours after single-dose administration and before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96 and 120 hours after last repeated-dose administration
metabolic clearance (CLM) for dapsone (DDS) | before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96 and 120 hours after single-dose administration and before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96 and 120 hours after last repeated-dose administration
rate of adverse events | participants will be followed for the duration of hospital stay (3 weeks) and up to 2 weeks after last study medication, an expected average of 5 weeks
Met-Hb | before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96 on study day 1 and 14 and additional once on study day 10 and 12
leucocytes | study day 12
erythrocytes | study day 12
hemoglobin | study day 12
hematocrit | study day 12
platelets | study day 12

CONTACTS AND LOCATIONS:
Overall Officials: Werner Siegmund, Prof, Principal Investigator — Department of Clinical Pharmacology
Locations (1):
- Department of Clinical Pharmacology, Ernst-Moritz-Arndt-University Greifswald, Greifswald, Mecklenburg-Vorpommern, Germany